CLINICAL TRIAL: NCT05094973
Title: Predictability of Distalization and Derotation of the Carriere Motion Appliance. A Clinical Study
Brief Title: Predictability of Distalization and Derotation of the Carriere Motion Appliance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Aldara Rosalía Nercellas Rodríguez, Principal Investigator, University of Salamanca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UniversidadSalamanca
Record Dates: First submitted 2021-09-28; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Dental Malocclusion
Keywords: Class II malocclusion; Carriere Motion Appliance; Distalization; Derotation
MeSH Terms: conditions — Malocclusion; Overbite

STUDY DESIGN:
Intervention Model Description: This study included 15 patients with Class II molar relationship and Class II canine relationship treated using Carriere Motion Appliance®.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Canine and molar distalization and molar derotation (Experimental): Evaluating the canine and molar distalization and molar derotation in dental Class II patients who where submitted to Carriere Motion Appliance® for a mean of 4 months.
  Interventions: Device: Carriere Motion Appliance®

INTERVENTIONS:
Device: Carriere Motion Appliance® — To analyze the distalization or distal tooth displacement and derotation angle produced by Carriere Motion Appliance® in a period of 4 months.

SUMMARY:
To analyze the distalization or distal tooth displacement and derotation angle produced by Carriere Motion Appliance® (CMA) by using a repeatable and reproducible measurement digital technique.

DETAILED DESCRIPTION:
15 patients with Class II molar and canine relationship were submitted to orthodontic treatment with CMA. All patients were exposed preoperatively (STL1) and postoperatively (STL2) to a digital impression and afterwards were uploaded into a specific cephalometric software to allow the automatic mesh networks alignment of the STL digital files. Subsequently, the distal tooth displacement of upper canines and first upper molars and also the derotation angle of first upper molars were measured. The repeatability and reproducibility were analyzed by Gage R&R statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Growing patients
* Late mixed dentition or permanent dentition
* Fully erupted definitive molars
* No history of previous orthodontic treatment
* Complete pre- and post-treatment records (digital study models)
* Dental Class II relationship.

Exclusion Criteria:

* Permanent dentition
* Adults
* Dental Class I, III

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Mean Canine Distalization | 4 months
  1.193 mm
Mean Molar Distalization | 4 months
  1.34 mm
Mean Molar Derotation | 4 months
  6.333º

CONTACTS AND LOCATIONS:
Overall Officials: Aldara Nercellas Rodríguez, Principal Investigator — University of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No